CLINICAL TRIAL: NCT03649581
Title: Investigation of Clinical, Cognitive and Neurophysiological Markers, Possibly Specific of Two Subforms of Psychotic Disorders
Brief Title: Investigation of Neurophysiological Markers, Possibly Specific of Two Subforms of Psychotic Disorders
Acronym: NeuroSplitsz
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7058
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient with schizophrenia and periodic catatonia (Experimental)
  Interventions: Other: compare the two groups of schizophrenic patients; Other: compare the two groups of schizophrenic patients versus volunteers
- patient with schizophrenia and hebephrenia (Experimental)
  Interventions: Other: compare the two groups of schizophrenic patients; Other: compare the two groups of schizophrenic patients versus volunteers
- healthy volunteers (Active Comparator)
  Interventions: Other: compare the two groups of schizophrenic patients; Other: compare the two groups of schizophrenic patients versus volunteers

INTERVENTIONS:
Other: compare the two groups of schizophrenic patients — Compare two groups of markers relating respectively to psychomotricity and affectivity in two subforms of schizophrenia: periodic catatonia and hebephrenia in order to highlight a possible double dissociation:
  1. abnormalities of markers related to affectivity in Hebephrenia (with preservation of these markers in periodic catatonia),
  2. abnormalities of markers related to psychomotricity in periodic catatonia (with markers of these tests in Hebephrenia).
Other: compare the two groups of schizophrenic patients versus volunteers — compare the results of the schizophrenic patient group with healthy volunteers

SUMMARY:
The current diagnostic criteria for schizophrenia and other psychotic disorders are relatively broad and lack precision. Therefore, distinct diseases may be grouped together under the same diagnostic category, although these diseases may differ according to their clinical expression, prognosis and perhaps their physiopathological causes.

We think that identifying subforms of psychotic disorders that are more homogeneous will better enable to understand their respective physiopathological causes and find personalized treatments.

This study will compare two subforms of psychotic disorders that have been clinically distinguished in the 1970s. These phenotypes have however not been validated yet using scientific investigations.

Using clinical assessments, cognitive evaluations and neurophysiological measures (fMRI) investigating the domains of affect and psychomotoricity , we expect that these two subforms will differ on their clinical, cognitive and neurophysiological characteristics, namely: hebephrenia will be associated with deficits on the affect markers , and respect psychomotoricity (catatonia scales, tests assessing movement planification) whereas the opposite pattern will be observed for periodic catatonia.

ELIGIBILITY:
Inclusion Criteria:

* for both patients and controls
* male or female willing to participate and who have signed up the legal document
* under the protection of health insurance for patients only
* schizophrenia or schizo-affective disorder according to the DSM-5 criteria
* periodic catatonia or hebephrenia accordin to WKL classification
* clinically stable for at least 2 months
* in or out patients for controls only
* no psychiatric history

Exclusion Criteria:

* for both patients and controls
* current severe or unstable somatic illness
* neurological history (epilepsia, brain injury, brain surgery…)
* current substance use disorder (DSM-5)
* current major depressive disorder (DSM-5)
* mental retardation (IQ < 70)
* pregnancy, breast feeding
* current legal control
* contra-indication for fMRI for controls only psychotropic intake during the last 3 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Index of affect | 6 months after inclusion
  Compare two groups of markers relating respectively to affectivity in two subforms of schizophrenia: periodic catatonia and hebephrenia in order to highlight a possible double dissociation
Index of psychomotoricity | 6 months after inclusion
  Compare two groups of markers relating to psychomotricity in two subforms of schizophrenia: periodic catatonia and hebephrenia in order to highlight a possible double dissociation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Psychiatrie I, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No